CLINICAL TRIAL: NCT03144232
Title: A Preliminary Investigation of Pre-Frontal Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Cannabis Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Gregory Sahlem, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 56294; K23DA043628 (NIH)
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There is a sham rTMS condition that will allow both participants and investigators to be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Experimental): 10 Hz rTMS applied to the left DLPFC
  Interventions: Device: Active rTMS
- Sham rTMS (Sham Comparator): Sham rTMS applied to the left DLPFC
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — rTMS will be delivered via a MagPro double blinded rTMS Research System (MagVenture, Denmark) with a Cool-B65 Butterfly Coil (a combined active and sham coil). We will use a standard resting motor threshold (rMT) determination to determine the TMS dose. Study-treatment will be delivered at 120% rMT. Each active rTMS study-treatment will consist of a total of 4000 pulses of 10Hz stimulation (5s-on,10s-off). Study-treatments will be delivered at the EEG coordinate for F3 (which approximates the left DLPFC), and will be found using the Beam-F3 method.
  Arms: Active rTMS
Device: Sham rTMS — Sham sessions will be delivered using an electronic sham system consisting of a coil that mimics the appearance and sound of rTMS, combined with a TENS device which produces a small electric shock mimicking the feeling of active rTMS. This type of sham has been demonstrated to be indistinguishable from active rTMS.
  Arms: Sham rTMS

SUMMARY:
This investigation will preliminarily determine if a course of high-frequency rTMS applied to the left dorsolateral prefrontal cortex, will reduce behavioral craving, and fMRI cue-reactivity in treatment-seeking cannabis use disordered participants.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to investigate if a course of excitatory DLPFC rTMS results in reduced cannabis behavioral craving in treatment-seeking individuals with CUD (Aim1). Additionally, the investigators seek to explore the mechanistic underpinnings of any observed effect, by collecting functional magnetic resonance imaging data during cannabis cue administration before and after the treatment course (Aim 2). These aims will be addressed through a nine-week, double-blind, randomized, sham-controlled study in which 72 treatment-seeking cannabis use disordered participants (36/group) will be given 20 sessions of either Active or Sham excitatory rTMS applied to the DLPFC. rTMS will be delivered over five weeks (2 sessions each day, two days each week). rTMS will be applied in conjunction with a validated three-session Motivational Enhancement Therapy (MET) behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Participants must be between the ages of 18 and 60.
3. Participants must meet DSM-5 criteria for at least moderate Cannabis Use Disorder, with use of at least 20 out of the last 28 days.
4. Participants must express a desire to quit cannabis.
5. Participants must have a Positive UDS for cannabis during their baseline visit (confirming they are regular users).

Exclusion Criteria:

1. Participants must not be pregnant or breastfeeding.
2. Participants must not meet moderate or severe use disorder of any other substance with the exception of Nicotine Use Disorder.
3. Participants must not be on any medications that have central nervous system effects.
4. Participants must not have a history of/or current psychotic disorder or bipolar disorder.
5. Participants must not have any other Axis I condition requiring current treatment and must have a HRSD24 ≤10 indicating no clinically relevant depressive symptoms.
6. Participants must not have a history of Dementia or other cognitive impairment.
7. Participants must not have active suicidal ideation, or a suicide attempt within the past 90 days.
8. Participants must not have any contraindications to receiving rTMS (e.g. metal implanted above the head, history of seizure, any known brain lesion).
9. Participants must not have any unstable general medical conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Repetitive Transcranial Magnetic Stimulation (rTMS): 10 Hz rTMS applied to the left dorsolateral prefrontal cortex (DLPFC).
Period: Overall Study
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham rTMS
Started | 37 | 35
Completed | 28 | 23
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham rTMS | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (9.9) | 30.7 (10.0) | 30.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 25 | 20 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 18 | 15 | 33
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 35 | 72

OUTCOME MEASURES:

1. Primary Outcome: Marijuana Craving Questionnaire-Short Form Score as a Measure of Behavioral Craving
Description: The investigators hypothesize that as compared to those participants receiving sham rTMS, those participants receiving active rTMS will have a reduced level of behavioral cannabis craving prior to their final rTMS session as compared to prior to their first rTMS session. The investigators will measure behavioral cannabis craving using the marijuana craving questionnaire. Score range: 12 to 84, higher scores represent more craving.
Time Frame: Baseline (pre) and Week-5 (post)
Population: All participants were included in the analysis using a mixed model, but the post-treatment mean and standard deviation only included available data (participants who completed treatment).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham rTMS
Number analyzed (Participants) | 37 | 35
score on a scale
  Pre | 45.8 (18.5) | 45.2 (16.3)
  Post: number analyzed (Participants) | 28 | 23
  Post | 27.7 (15.1) | 22.6 (11.1)

2. Primary Outcome: Cue Reactivity
Description: The investigators hypothesize that as compared to those participants receiving sham rTMS, those participants receiving active rTMS will have a reduced BOLD response in reward structures (dorsal striatum, ventral striatum, and anterior consulate cortex) during a validated cue-reactivity fMRI paradigm prior to their final rTMS session as compared to prior to their first rTMS session (change score). The following beta scores represent the change score (post-pre) in scans in the drug stimuli minus neutral stimuli subtraction map. Generally, more activation (a positive score) represents more cannabis image cue-reactivity, and the reported range represents standard units as output in the fMRI.
Time Frame: Baseline (pre) and Week-5 (post)
Population: Participants with data at both pre and post time-points were included in the analysis.
Measure: Mean (Standard Deviation); unit: BOLD signal change
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham rTMS
Number analyzed (Participants) | 23 | 17
BOLD signal change
  Ventral Striatum | 0.010 (0.164) | -0.025 (0.138)
  Dorsal Striatum | -0.013 (0.106) | -0.022 (0.122)
  Anterior Cingulate Cortex | 0.003 (0.167) | -0.015 (0.125)

3. Secondary Outcome: Abstinence
Description: Number of weeks (out of a total of 4 possible), in the follow-up period, where participants were abstinent from cannabis. Missing data was conservatively assumed to be non-abstinant. More weeks of abstinence is more favourable
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham rTMS
Number analyzed (Participants) | 37 | 35
weeks | .62 (1.21) | .37 (.77)

ADVERSE EVENTS:
Time Frame: 9-weeks
Arm/Group | Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 16/37 | 7/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Repetitive Transcranial Magnetic Stimulation (rTMS) (N=37) | Sham rTMS (N=35)
Headache (Nervous system disorders) | 10 | 4
Fatigue (Nervous system disorders) | 6 | 3
Eye twitch (Eye disorders) | 1 | 0
Jaw Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Site discomfort (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Mood Swings (Psychiatric disorders) | 0 | 1
Hand numbness (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Amendment 1.2 (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT03144232/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Final Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03144232/SAP_001.pdf